CLINICAL TRIAL: NCT05800704
Title: Randomized, Controlled, Double-blind, Parallel, Multicentric Study to Investigate Support of the Colonization Resistance of the Gut Microbiota with the Synbiotic Food Supplement Nagasin® After Disturbance by Antimicrobial Treatment
Brief Title: Support of Colonization Resistance of the Gut Microbiota with the Synbiotic Food Supplement Nagasin®
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Insel Gruppe AG, University Hospital Bern (Other); Stadtspital Zürich (Other); Kantonsspital Winterthur KSW (Other); Luzerner Kantonsspital (Other); Cantonal Hosptal, Baselland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: BASEC 2022-01318
Record Dates: First submitted 2023-03-23; First posted 2023-04-06 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: C. Difficile Enteritis
Keywords: Gut microbiota; Colonization resistance; Gut microbiota dysbiosis
MeSH Terms: interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nagasin® (Experimental): consumption of Nagasin® (synbiotic food supplement) once per day for four weeks
  Interventions: Dietary Supplement: Nagasin
- Comparator (Placebo Comparator): consumption of the comparator (maltodextrin) once per day for four weeks
  Interventions: Dietary Supplement: maltodextrin

INTERVENTIONS:
Dietary Supplement: Nagasin — Lactobacillus, Lactococcus and Bifidobacteria strains with antimicrobial effect against C. difficile
  Arms: Nagasin®
Dietary Supplement: maltodextrin — maltodextrin (placebo comparator)
  Arms: Comparator

SUMMARY:
Double blind, placebo-controlled, parallel, multicentric trial to investigat whether Nagasin® can support the colonization resistance against C.difficile.

DETAILED DESCRIPTION:
The aim of this randomized, controlled, double-blind, parallel, multicentric trial is to investigate wether the synbiotic food supplement Nagasin® can support the colonization resistance of the gut microbiota after disturbance by antimicrobial treatment.

The main question is whether Nagasin® can prevent any increase in abundance of C.difficile within the first four weeks after antimicrobial treatment for a C. difficile infection.

Participants will receive Nagasin® or the comparator as a food supplement during the first four weeks after antimicrobial treatment for a C. difficile episode.

ELIGIBILITY:
Inclusion Criteria:

* C. difficile infection (CDI) diagnosis
* antimicrobial treatment (e.g. metronidazole, vancomycin or fidaxomicin) for C. difficile infection at ICF
* Written informed consent by the participant after information about the research project

Exclusion Criteria:

* total parenteral nutrition
* insulin-dependent (type 1) diabetes
* severe disease defined as any of the following:

  * White blood cell count (WBC) > 30,000 or < 1000 cells/mm3
  * Neutropenia < 500 x 10^9 per liter
  * Intensive care unit (ICU) patient at time C. difficile infection diagnosed
  * In case no hematology values are available, presence of severe can be evaluated by the local principal investigator or his designee
* is severely immunocompromised as defined by any of the following:

  * active malignancy receiving severe immunosuppressive chemotherapy with subsequent leukopenia (as defined above)
  * long-term systemic steroid therapy ≥ 30 mg / d
  * recipients of stem cell transfer (≤ 12 months)
  * severe inborn immune deficiency or severe immunosuppressive therapy as evaluated by the investigator
  * HIV patients with low CD4+ cell count (< 200 x 10^9 per liter)
  * Inflammatory bowel disease patients if:
  * severe ulcerative colitis (classified as endoscopic Mayo = 3 (max. 30 days old) or as evaluated by investigator)
  * Severe Crohn's disease with acute penetrating complication (abscess and/or actively draining fistulae) or as evaluated by investigator
  * Liver cirrhosis (classified as Child C) with clinically significant portal hypertension and/or low thrombocyte count (20 × 10^9 per liter)
* Acute pancreatitis
* prosthetic heart valves or endocarditis
* consumption of other high-dose (>10^10 cfu/dose) probiotic products during the study period.
* Inability to understand and follow study procedures
* prosthetic heart valves or endocarditis
* consumption of other high-dose (>10^10 cfu/dose) probiotic products during the study period.
* Inability to understand and follow study procedures

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2023-03-10 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
C. difficile relative abundance | at 1, 2 and 4 weeks after completion of antimicrobial treatment for CDI
  any change of C. difficile relative abundance during the first four weeks after antimicrobial treatment for CDI.

SECONDARY OUTCOMES:
Gut microbiota | at 1, 2, 4 and 8 weeks after completion of antimicrobial treatment for CDI
  Gut microbiota diversity and taxonomic composition
Abundance of antibiotic diarrhea associated pathogens | at 1, 2, 4 and 8 weeks after completion of antimicrobial treatment for CDI
  Abundance of other pathogens that are involved in antibiotic associated diarrhea e.g. S. aureus and K. oxytoca
C. difficile toxins | at 1, 2, 4 and 8 weeks after completion of antimicrobial treatment for CDI
  Presence and amount of C. difficile toxins
Toxin forming C. difficile strains | at 1, 2, 4 and 8 weeks after completion of antimicrobial treatment for CDI
  Presence of toxin forming C. difficile strains

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle M Frey-Wagner, PhD, Study Chair — University or Zurich, Institute of Medical Microbiology
Locations (6):
- Switzerland (6):
  - Kantonsspital Baselland, Liestal, Basel-Landschaft
  - Inselspital Bern, Bern, Canton of Bern
  - Luzerner Kantonsspital, Lucerne, Canton of Lucerne
  - Kantonsspital Winterthur, Winterthur, Canton of Zurich
  - Stadtspital Zürich, Zurich, Canton of Zurich
  - University Hospital Zurich, Zurich, Canton of Zurich

IPD SHARING:
Plan to Share IPD: No